CLINICAL TRIAL: NCT01995175
Title: A Prospective, Epidemiological Study to Assess the Disease Burden of RSV Associated, Suspected LRTIs From 0 to 2 Years and Population Attributable Risk Percent of RSV LRTI on the Development of Recurrent Wheeze and Asthma From 0 to 6 Years
Brief Title: A Prospective, Epidemiological Study to Assess the Disease Burden of Respiratory Syncytial Virus Associated, Suspected Lower Respiratory Tract Infections in Newborns, From 0 to 2 Years of Age and Risk of Development of Wheeze and Asthma From 0 to 6 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200150
Record Dates: First submitted 2013-11-07; First posted 2013-11-26 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Syncytial Virus
Keywords: Asthma; Respiratory Syncytial virus; Cohort study; Quarterly phone contacts; Wheeze; New born; Lower Respiratory Tract Infection
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Blood Specimen Collection

ARMS (1):
- Overall Group (Other): Newborn subjects followed up for Lower Respiratory Tract Infections (LRTI) symptoms from birth until they are 2 years of age and for incidence of wheeze and asthma up to 6 years of age.
  Interventions: Procedure: Nasal swab sampling; Procedure: Blood sampling; Other: Diary cards

INTERVENTIONS:
Procedure: Nasal swab sampling — Nasal swab samples will be collected from subjects at each examination visit, if they develop respiratory tract infection symptoms with difficulty in breathing and are called for an examination visit in the study.
Procedure: Blood sampling — A single blood sample will be collected from a sub-cohort consisting of the first 2000 enrolled subjects when they are either 2, 4, 6, 12, 18 or 24 months old.
Other: Diary cards — Diary cards will be provided to parents or LARs of the subjects to record RTI/LRTI, wheeze and asthma symptoms.

SUMMARY:
The purpose of this study is to assess the incidence and associated healthcare utilization of RSV-associated, suspected LRTI in a general population of infants from birth up to 2 years of age, and also to assess the accuracy of a newly developed LRTI case definition and severity scale compared to two existing definitions. The study will also assess the population attributable risk percent of RSV LRTI on the development of wheeze and asthma from 0 to 6 years of age.

DETAILED DESCRIPTION:
New born infants from various countries over the world will be followed up for up to two years for the occurrence of Lower Respiratory Tract Infections. Through active and passive surveillance, any suspected case will be identified, assessed during an examination visit and followed up until completion through a diary card. Full symptomology will be assessed during the examination visit. The disease course and all healthcare utilization will be subsequently collected through a two-week diary card and contact with ay healthcare providers involved in management of the disease. RSV detection will occur through quantitative PCR of collected nasal swabs. A baseline cord blood serum sample of all subjects and a follow-up blood serum sample from a sub-cohort will also be collected to assess antibody levels at various points in time and in relation to risk of RSV LRTI.

For extension period, pertaining to wheeze and asthma (Epoch 002): Subjects' parent(s)/LAR(s) will be asked to re-consent and subjects will be followed up through quarterly contacts up to the age of 6 years. Data collection will also occur from medical charts retrospectively for those who have a gap period between the end of the primary study and providing re-consent for the extension. The extension involves enrolment visit (at 2nd birthday [on completion of primary study or as soon as possible thereafter]) and quarterly surveillance contacts.

ELIGIBILITY:
Inclusion Criteria:

Before birth:

* Subject whose parent(s)/Legally Acceptable Representative(s) (LARs), in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent (including consent to obtain a cord blood sample at birth) obtained from the parent(s)/LAR(s) of the subject.

After Birth:

* Subject for whom updated and re-signed informed consent and confirmation of eligibility is available not later than 5 working days after birth.
* Cord blood sample collection of at least 3 mL, at birth.

For extension period:

* Subject is enrolled at a study site that is participating in the extension period follow-up.
* Subject whose parent(s)/LAR(s), in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent (or witnessed thumb printed consent in case of an illiterate subject) obtained from the parent(s)/LAR(s) of the subject.
* Previous participation in the primary study (from birth up to the age of 2 years).

Exclusion Criteria:

Before birth:

* Subject expected to become Child in care
* Subjects whose parent(s)/LAR(s) are below the age of 18 or the legal consenting age of the respective country if this is higher.

After Birth:

* Child in care
* Newborn with a gestational age of less than 28 weeks.
* Subjects with any congenital condition that will require an expected postnatal stay in hospital of more than 12 consecutive weeks.
* Subjects with major congenital defects or serious chronic illness limiting life expectancy to less than 5 years.
* Subjects with any confirmed or suspected immunosuppressive or immunodeficient condition (including positive infection with human immunodeficiency virus [HIV]), based on medical history, physical examination or positive test result.

For extension period:

• Child in care.

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2409 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (8):
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Seattle, Washington
- Argentina (2):
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Río Cuarto
- GSK Investigational Site, Dhaka, Bangladesh
- GSK Investigational Site, Halifax, Nova Scotia, Canada
- Finland (4):
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
- GSK Investigational Site, San Pedro Sula, Honduras
- GSK Investigational Site, Soweto, Gauteng, South Africa
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Pathum Thani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madhi SA, Ceballos A, Cousin L, Domachowske JB, Langley JM, Lu E, Puthanakit T, Ramet M, Tan A, Zaman K, Anspach B, Bueso A, Cinconze E, Colas JA, D'Andrea U, Dieussaert I, Englund JA, Gandhi S, Jose L, Kim JH, Klein NP, Laajalahti O, Mithani R, Ota MOC, Pinto M, Silas P, Stoszek SK, Tangsathapornpong A, Teeratakulpisarn J, Virta M, Cohen RA. Population Attributable Risk of Wheeze in 2-<6-Year-old Children, Following a Respiratory Syncytial Virus Lower Respiratory Tract Infection in The First 2 Years of Life. Pediatr Infect Dis J. 2025 May 1;44(5):379-386. doi: 10.1097/INF.0000000000004447. Epub 2024 Jul 1. PMID 38985986
- [Derived] Englund JA, Cohen RA, Bianco V, Domachowske JB, Langley JM, Madhi SA, Zaman K, Bueso A, Ceballos A, Cousin L, Gandhi S, Gruselle O, Jose L, Klein NP, Koen A, Puthanakit T, Shi M, Silas P, Tangsathapornpong A, Teeratakulpisarn J, Vesikari T, Haars G, Leach A, Stoszek SK, Dieussaert I. Evaluation of Clinical Case Definitions for Respiratory Syncytial Virus Lower Respiratory Tract Infection in Young Children. J Pediatric Infect Dis Soc. 2023 May 31;12(5):273-281. doi: 10.1093/jpids/piad028. PMID 37142551
- [Derived] Langley JM, Bianco V, Domachowske JB, Madhi SA, Stoszek SK, Zaman K, Bueso A, Ceballos A, Cousin L, D'Andrea U, Dieussaert I, Englund JA, Gandhi S, Gruselle O, Haars G, Jose L, Klein NP, Leach A, Maleux K, Nguyen TLA, Puthanakit T, Silas P, Tangsathapornpong A, Teeratakulpisarn J, Vesikari T, Cohen RA. Incidence of Respiratory Syncytial Virus Lower Respiratory Tract Infections During the First 2 Years of Life: A Prospective Study Across Diverse Global Settings. J Infect Dis. 2022 Aug 26;226(3):374-385. doi: 10.1093/infdis/jiac227. PMID 35668702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2409 subjects were enrolled in the primary study and followed-up from birth up to 2 years of age (Period 1 - from 0 up to 2 years of age). 1395 subjects from primary study were enrolled in the extension study and followed-up from 2 up to 6 years of age (Period 2 - from 2 up to 6 years of age).
Pre-assignment Details: Out of 2409 subjects enrolled in the primary study, 7 subjects did not sign the re-consent for study participation after delivery (birth), leaving 2402 subjects enrolled. 1 subject was excluded due to protocol violation, hence 2401 subjects formed the Per Protocol Set-Primary Study. Out of 2148 subjects who completed the primary study, 10 subjects were excluded due to invalid ICF/fraudulent data, 743 did not further participate, and therefore, 1395 subjects were enrolled in the extension study.
Period: Period 1 - From 0 up to 2 Years of Age
Arm/Group | Overall Group
Started | 2401
Completed (Completed=Number of subjects that completed the primary study) | 2148
Not Completed | 253
Not completed — Withdrawal by Subject | 35
Not completed — Lost to Follow-up | 102
Not completed — Other | 67
Not completed — Migrated / moved from the study area | 49
Period: Period 2 - From 2 up to 6 Years of Age
Arm/Group | Overall Group
Started | 1395 (Out of 2148 subjects who completed the primary study, 10 subjects were excluded from the extension study due to invalid informed consent form (ICF) or fraudulent data, and 743 subjects were at a site that did not participate, or they did not consent to participate in the extension study.)
Completed | 1338
Not Completed | 57
Not completed — Other | 21
Not completed — Lost to Follow-up | 22
Not completed — Migrated/moved from the study area | 6
Not completed — Consent withdrawal, not due to a Serious Adverse Event | 7
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Age, Customized [Count of Participants; unit: Participants] — Period 1 - From 0 up to 2 years of age
  Participants
    Gestational age at birth ≤28 weeks | 0
    Gestational age at birth 29-32 weeks | 26
    Gestational age at birth 33-36 weeks | 154
    Gestational age at birth ≥37 weeks | 2221
Age, Customized [Count of Participants; unit: Participants] — Period 2 - From 2 up to 6 years of age Population: Period 2 - From 2 up to 6 years of age
  Participants
    24 to 36 months of age: number analyzed (Participants) | 1395
    24 to 36 months of age | 1395
Sex/Gender, Customized [Count of Participants; unit: Participants] — Period 1 - From 0 up to 2 years of age
  Participants
    Male | 704
    Female | 729
    Missing | 968
Sex/Gender, Customized [Count of Participants; unit: Participants] — Period 2 - From 2 up to 6 years of age Population: Period 2 - From 2 up to 6 years of age
  Participants
    Male: number analyzed (Participants) | 1395
    Male | 687
    Female: number analyzed (Participants) | 1395
    Female | 708
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Period 1 - From 0 up to 2 years of age
  Participants
    Geographic ancestry: African Heritage / African American | 632
    Geographic ancestry: American Indian or Alaskan Native | 7
    Geographic ancestry: Asian - Central/South Asian Heritage | 5
    Geographic ancestry: Asian - East Asian Heritage | 4
    Geographic ancestry: Asian - Japanese Heritage | 1
    Geographic ancestry: Asian - South East Asian Heritage | 435
    Geographic ancestry: Latino/Mestizo | 303
    Geographic ancestry: Native Hawaiian or Other Pacific Islander | 3
    Geographic ancestry: White - Arabic / North African Heritage | 6
    Geographic ancestry: White - Caucasian / European Heritage | 888
    Geographic ancestry: Not specified | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Period 2 - From 2 up to 6 years of age Population: Period 2 - From 2 up to 6 years of age
  Participants
    Geographic ancestry: number analyzed (Participants) | 1395
    Geographic ancestry: African Heritage / African American | 386
    Geographic ancestry: American Indian or Alaskan Native | 4
    Geographic ancestry: Asian - Central/South Asian Heritage | 3
    Geographic ancestry: Asian - East Asian Heritage | 4
    Geographic ancestry: Asian - Japanese Heritage | 1
    Geographic ancestry: Asian - South East Asian Heritage | 271
    Geographic ancestry: Latino/Mestizo | 103
    Geographic ancestry: Native Hawaiian or Other Pacific Islander | 2
    Geographic ancestry: White - Arabic / North African Heritage | 2
    Geographic ancestry: White - Caucasian / European Heritage | 549
    Geographic ancestry: Not specified | 70

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates of First Episode of Respiratory Syncytial Virus (RSV) Respiratory Tract Infection (RTI) [Period 1]
Description: The incidence rate was calculated by dividing the number of subjects reporting first episode over the follow-up period, to the total person-years. Detection of the RSV-infection was performed by reverse transcription quantitative real time polymerase chain reaction (RT-qPCR ) assay on ribonucleic acids (RNA) extracted from nasal swabs. Number of suspected RSV RTI cases were tabulated.
Time Frame: From birth up to 2 years of age
Population: The analysis was performed on the Per Protocol Set (PPS) which included all subjects enrolled in the primary study meeting all eligibility criteria up to the time of their censoring, either at completion of primary study or prematurely as drop-out (e.g., withdrawn consent, lost-to-follow-up).
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Cases per 100 person-years | 7.93 [7.10 to 8.84]

2. Primary Outcome: Number of Subjects Hospitalized for RSV [Period 1]
Description: Healthcare utilization included primary, secondary and tertiary care settings such as self-care with Over-The-Counter [OTC] drugs, general practitioner [GP] visits, emergency room [ER] visits, hospital visits, etc. Note: This outcome measure presents results only for the more severe events of healthcare utilization - RSV hospitalization. Results for other causes (non-RSV) hospitalization and healthcare utilization for other settings were not calculated, as data were not available.
Time Frame: From birth up to 2 years of age
Population: The analysis was performed on the Per Protocol Set (PPS) which included all subjects enrolled in the primary cohort study meeting all eligibility criteria up to the time of their censoring, either at completion of epoch 1 or prematurely as drop-out (e.g., withdrawn consent, lost-to-follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Participants | 31

3. Primary Outcome: Incidence Rates of RSV Lower Respiratory Tract Infection (LRTI) or Severe LRTI as Defined by the LRTI Case Definition and Severity Scale [Period 1]
Description: The incidence rate was calculated by dividing the number of subjects reporting first episodes over the follow-up period, to the total person-years. LRTI Case definition by WHO (Modjarrad 2015): LRTI is diagnosed when a child <5 years presents with cough and/or difficulty in breathing has the following symptoms: Fast breathing, (>60 per minute in a child <2 m, >50 per minute in a child 2 to 11 m and >40 per minute in a child 12 to 59 m) or Oxygen saturation <95% by pulse oximetry.
  Severe LRTI is diagnosed when an infant with RSV LRTI has oxygen saturation<93% or lower chest wall drawing.
Time Frame: From birth up to 2 years of age
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Cases per 100 person-years
  WHO RSV LRTI | 4.75 [4.13 to 5.45]
  WHO RSV severe LRTI | 1.53 [1.19 to 1.94]

4. Primary Outcome: Number of RSV LRTI or Severe LRTI Episodes as Defined by the GlaxoSmithKline (GSK) LRTI Case Definition [Period 1]
Description: LRTI Case definition by GSK: LRTI is diagnosed when a child <5 years presents with cough or runny or blocked nose and oxygen saturation <95% with a respiratory rate ≥ 60/minute (< 2 months of age); ≥ 50/minute (2 to 11 months of age); ≥ 40/minute (12 to 24 months of age) and has RSV infection, confirmed on nasal swab positive for RSV A or B by quantitative polymerase chain reaction (qPCR).
  Severe LRTI case definition by GSK: Child with LRTI and oxygen saturation < 92%, OR Difficulty breathing leading to: Irritability/agitation, or Lethargy/sleepiness, or Severe chest indrawing, or Reduced/no vocalization, or Apnoea > 20 sec, or Cyanosis, or Stop feeding well/dehydration.
Time Frame: From birth up to 2 years of age
Population: The analysis was performed on the RSV LRTI or severe LRTI episodes collected from subjects in the PPS.
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Number analyzed (Episodes) | 1652
Episodes
  GSK RSV LRTI episodes | 227
  GSK severe RSV LRTI episodes | 145

5. Primary Outcome: Number of RSV LRTI or Severe LRTI Episodes as Defined by the Existing Comparator LRTI Case Definition (WHO [Modjarrad 2015]) [Period 1]
Description: LRTI is diagnosed when a child <5 years presents with cough and/or difficulty in breathing has the following symptoms: Fast breathing, (>60 per minute in a child <2 m, >50 per minute in a child 2 to 11 m and >40 per minute in a child 12 to 59 m) or Oxygen saturation <95% by pulse oximetry. Severe LRTI is diagnosed when a child has LRTI and Oxygen saturation <93% by pulse oximetry and/or lower chest wall in-drawing.
Time Frame: From birth up to 2 years of age
Population: The analysis was performed on the suspected RSV LRTI or severe LRTI episodes reported by subjects in the PPS.
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Number analyzed (Episodes) | 1652
Episodes
  WHO RSV LRTI episodes | 227
  WHO severe RSV LRTI episodes | 73

6. Primary Outcome: Number of RSV LRTI or Severe LRTI Episodes as Defined by the Existing Comparator LRTI Case Definition (Nokes et al.) [Period 1]
Description: LRTI is diagnosed when a child has a history of acute cough or difficulty in breathing and greater than or equal to (≥) 1 of the following: Fast breathing for age (≥ 60 breaths/minimum if the child is < 2 m ≥ 50 breaths/minimum if the child is 2-11 m). Indrawing, or Low oxygen saturation (< 90%) by pulse oximetry or inability to feed (prostration or unconsciousness), when accompanied by a clinical diagnosis of LRTI or bronchiolitis. Severe LRTI is diagnosed when a child has Indrawing, or Low oxygen saturation (< 90%) by pulse oximetry or inability to feed (prostration or unconsciousness), when accompanied by a clinical diagnosis of LRTI or bronchiolitis.
Time Frame: From birth up to 2 years of age
Population: The analysis was performed on the suspected RSV LRTI or severe LRTI episodes collected from subjects in the PPS.
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Number analyzed (Episodes) | 1652
Episodes
  Nokes et al. RSV LRTI episodes | 226
  Nokes et al. severe RSV LRTI episodes | 67

7. Secondary Outcome: Levels of RSV-A and B Neutralizing Antibodies in the Cord Blood [Period 1]
Description: Levels of RSV A and B neutralizing antibodies were expressed as Geometric Mean Titers (GMTs) and the cut off for the neutralization assay was 8 End Point Dilution 60 percent (ED60) for RSV-A antibodies and 6 ED60 for RSV-B antibodies. Infant baseline blood sample serum was tested for detection of RSV neutralizing antibodies level.
Time Frame: At birth (Month 0)
Population: The analysis was performed on the Per Protocol Set (PPS) which included all subjects enrolled in the primary study meeting all eligibility criteria and for whom immunogenicity data were available at the time point considered and for the measured antibody.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Overall Group
Number analyzed (Participants) | 2390
Titers
  RSV-A at Month 0 (Overall) | 251.21 [241.31 to 261.51]
  RSV-B at Month 0 (Overall): number analyzed (Participants) | 2355
  RSV-B at Month 0 (Overall) | 327.05 [315.17 to 339.38]

8. Secondary Outcome: Levels of RSV-A and B Neutralizing Antibodies in the Blood Serum [Period 1]
Description: Levels of RSV A and B neutralizing antibodies were expressed as GMTs and the cut off for the neutralization assay was 8 End Point Dilution 60 percent (ED60) for RSV-A antibodies and 6 ED60 for RSV-B antibodies. Infant blood sample serum was tested for RSV neutralizing antibodies level detection.
Time Frame: At 2, 4, 6, 12, 18 and 24 months of age
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Overall Group
Number analyzed (Participants) | 1384
Titers
  RSV-A at Month 2: number analyzed (Participants) | 174
  RSV-A at Month 2 | 77.92 [67.70 to 89.68]
  RSV-A at Month 4: number analyzed (Participants) | 176
  RSV-A at Month 4 | 31.25 [26.79 to 36.46]
  RSV-A at Month 6: number analyzed (Participants) | 184
  RSV-A at Month 6 | 13.91 [11.96 to 16.17]
  RSV-A at Month 12: number analyzed (Participants) | 231
  RSV-A at Month 12 | 14.30 [11.83 to 17.29]
  RSV-A at Month 18: number analyzed (Participants) | 306
  RSV-A at Month 18 | 22.41 [18.30 to 27.44]
  RSV-A at Month 24: number analyzed (Participants) | 313
  RSV-A at Month 24 | 46.32 [37.85 to 56.67]
  RSV-B at Month 2: number analyzed (Participants) | 173
  RSV-B at Month 2 | 104.29 [91.17 to 119.31]
  RSV-B at Month 4: number analyzed (Participants) | 168
  RSV-B at Month 4 | 50.59 [44.13 to 58.00]
  RSV-B at Month 6: number analyzed (Participants) | 176
  RSV-B at Month 6 | 30.25 [25.82 to 35.45]
  RSV-B at Month 12: number analyzed (Participants) | 223
  RSV-B at Month 12 | 20.45 [16.08 to 26.02]
  RSV-B at Month 18: number analyzed (Participants) | 281
  RSV-B at Month 18 | 31.32 [24.33 to 40.33]
  RSV-B at Month 24: number analyzed (Participants) | 302
  RSV-B at Month 24 | 59.89 [47.45 to 75.61]

9. Secondary Outcome: GMTs of RSV A and B Neutralizing Antibodies in the Cord Blood by Subjects Classified According to Non-overlapping Disease Severity Categories [Period 1]
Description: The association between RSV LRTI, RSV severe LRTI and RSV A and B neutralizing antibodies were assessed by calculating the GMTs of RSV A and B neutralizing antibodies in the cord blood by subjects classified according to non-overlapping disease severity categories: Non case (defined as subject not reporting RSV LRTI or RSV severe LRTI), WHO RSV LRTI (excluding WHO RSV severe LRTI) and WHO RSV severe LRTI.
Time Frame: At Month 0
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Overall Group
Number analyzed (Participants) | 2390
Titers
  Non case- RSV A: number analyzed (Participants) | 2349
  Non case- RSV A | 252.47 [242.41 to 262.94]
  WHO RSV LRTI- RSV A: number analyzed (Participants) | 21
  WHO RSV LRTI- RSV A | 213.24 [153.23 to 296.77]
  WHO RSV Severe LRTI- RSV A: number analyzed (Participants) | 20
  WHO RSV Severe LRTI- RSV A | 165.80 [110.78 to 248.14]
  Non Case- RSV B: number analyzed (Participants) | 2314
  Non Case- RSV B | 328.18 [316.12 to 340.71]
  RSV LRTI- RSV A: number analyzed (Participants) | 21
  RSV LRTI- RSV A | 259.18 [182.97 to 367.12]
  RSV severe LRTI- RSV A: number analyzed (Participants) | 20
  RSV severe LRTI- RSV A | 279.69 [205.47 to 380.73]

10. Secondary Outcome: GMTs of RSV A and B Neutralizing Antibodies by Subjects Classified According to Non-overlapping Disease Severity Categories [Period 1]
Description: The association between RSV LRTI, RSV severe LRTI and RSV A and B neutralizing antibodies were assessed by calculating the GMTs of RSV A and B neutralizing antibodies by subjects classified according to non-overlapping disease severity categories: Non case (defined as subject not reporting RSV LRTI or RSV severe LRTI), RSV LTRI and RSV severe LRTI.
Time Frame: During the first 6 months of life
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Overall Group
Number analyzed (Participants) | 2305
Titers
  Non case- RSV A: number analyzed (Participants) | 2304
  Non case- RSV A | 254.08 [243.84 to 264.76]
  WHO RSV LRTI- RSV A: number analyzed (Participants) | 47
  WHO RSV LRTI- RSV A | 193.34 [154.08 to 242.60]
  WHO RSV Severe LRTI- RSV A: number analyzed (Participants) | 38
  WHO RSV Severe LRTI- RSV A | 174.09 [132.41 to 228.89]
  Non Case- RSV B: number analyzed (Participants) | 2271
  Non Case- RSV B | 327.83 [315.62 to 340.51]
  RSV LRTI- RSV B: number analyzed (Participants) | 47
  RSV LRTI- RSV B | 276.52 [222.70 to 343.36]
  RSV severe LRTI- RSV B: number analyzed (Participants) | 37
  RSV severe LRTI- RSV B | 349.53 [279.11 to 437.71]

11. Secondary Outcome: Number of WHO LRTI Episodes by Age Categories [Period 1]
Description: LRTI refers to Child with RTI AND Blood Oxygen Saturation (SaO2) lower than (<) 95 percent (%), OR respiratory rate (RR) increase: higher than (>) 60/min < 2 months (m) of age; > 50/min 2-11m of age, 40/min 12-24m of age. Severe LRTI refers to Child with LRTI AND SaO2 < 92%, OR Difficulty breathing leading to: Irritability/agitation, OR Lethargy/sleepiness, OR Severe chest indrawing, OR Reduced/no vocalization, OR Apnoea > 20 sec, OR Cyanosis, OR Stop feeding well/dehydration. The number of WHO LRTI cases were assessed for the following age groups: 0-2, 3-5, 6-11 and 12-23 months of age. Occurrence of LRTI/severe LRTI cases as classified by the LRTI case definitions and severity scale, was not limited to the subgroups of subjects recruited from Months 1-6 and 13-18 but was provided for subjects in all age intervals: 0-2 months, 3-5 months, 6-11 months and 12-23 months.
Time Frame: From birth up to 2 years of life
Population: The analysis was performed on the WHO LRTI episodes collected from subjects in the PPS.
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Number analyzed (Episodes) | 1012
Episodes
  0-2 Months | 110
  3-5 Months | 210
  6-11 Months | 276
  12-23 Months | 416

12. Secondary Outcome: Number of WHO Severe LRTI Cases by Age Categories [Period 1]
Description: LRTI refers to Child with RTI AND Blood Oxygen Saturation (SaO2) lower than (<) 95 percent (%), OR respiratory rate (RR) increase: higher than (>) 60/min < 2 months (m) of age; > 50/min 2-11m of age, 40/min 12-24m of age. Severe LRTI refers to Child with LRTI AND SaO2 < 92%, OR Difficulty breathing leading to: Irritability/agitation, OR Lethargy/sleepiness, OR Severe chest indrawing, OR Reduced/no vocalization, OR Apnoea > 20 sec, OR Cyanosis, OR Stop feeding well/dehydration. The number of WHO severe LRTI cases were assessed for the following age groups: 0-2, 3-5, 6-11 and 12-23 months of age.
Time Frame: From birth up to 2 years of life
Population: The analysis was performed on WHO severe LRTI episodes collected from subjects in the PPS.
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Arm/Group | Overall Group
Number analyzed (Participants) | 2401
Number analyzed (Episodes) | 259
Episodes
  0-2 Months | 45
  3-5 Months | 67
  6-11 Months | 62
  12-23 Months | 85

13. Secondary Outcome: Incidence Rates of First Episode of Medically Attended Wheeze [Period 2]
Description: The incidence rate was calculated by dividing the number of subjects reporting first episode of medically attended wheeze over the follow-up period, to the total person-years. Medically attended wheeze = an episode of health care provider confirmed wheeze. Medically attended wheeze, in the extension phase, was collected via a history from parents solicited by contact every 3 months, which was supplemented by the review of routine medical records or contact with health care provider. Incidence rate was assessed for the following categories: All subjects, Non-case (defined as subject not reporting RSV LRTI or RSV severe LRTI) and WHO RSV LRTI.
Time Frame: From 2 years of age up to 6 years of age
Population: The analysis was performed on the PPS extension study, which included all subjects who met the eligibility criteria for the extension study up to the time of their censoring, either at study completion or prematurely as drop-out.
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Overall Group
Number analyzed (Participants) | 1395
Cases per 100 person-years
  All Subjects | 3.79 [3.27 to 4.37]
  Non-case: number analyzed (Participants) | 1269
  Non-case | 3.28 [2.78 to 3.85]
  WHO RSV LRTI: number analyzed (Participants) | 126
  WHO RSV LRTI | 9.82 [6.95 to 13.47]

14. Secondary Outcome: Incidence Rates of First Episode of Wheeze or Asthma Requiring Hospital Admission [Period 2]
Description: The incidence rate was calculated by dividing the number of subjects reporting first episode of wheeze or asthma requiring hospital admission over the follow-up period, to the total person-years. Wheeze or asthma requiring hospital admission = an episode of health care provider confirmed wheeze or asthma requiring hospital admission. Wheeze or asthma requiring hospital admission, in the extension phase, was collected via a history from parents, which was supplemented by the review of routine medical records or contact with health care provider. Incidence rate was assessed for the following categories: All subjects, Non-case (defined as subject not reporting RSV LRTI or RSV severe LRTI) and WHO RSV LRTI.
Time Frame: From 2 years of age up to 6 years of age
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Overall Group
Number analyzed (Participants) | 1395
Cases per 100 person-years
  All subjects | 0.35 [0.21 to 0.55]
  Non-case: number analyzed (Participants) | 1269
  Non-case | 0.30 [0.17 to 0.50]
  WHO RSV LRTI: number analyzed (Participants) | 126
  WHO RSV LRTI | 0.82 [0.22 to 2.09]

15. Secondary Outcome: Incidence Rates of First Episode of Reported Wheeze With Use of Any Medication [Period 2]
Description: The incidence rate was calculated by dividing the number of subjects reporting first episode of reported wheeze with use of any medication over the follow-up period, to the total person-years. Reported wheeze = parents report a whistling sound associated with labored breathing. Prescription of medications for wheeze, in the extension phase, was collected via a specific request for relevant medication from parents, which was supplemented by the review of routine medical records or contact with health care provider. Incidence rate was assessed for the following categories: All subjects, Non-case (defined as subject not reporting RSV LRTI or RSV severe LRTI) and WHO RSV LRTI.
Time Frame: From 2 years of age up to 6 years of age
Population: The analysis was performed on the PPS extension study which included all subjects who met the eligibility criteria for the extension study up to the time of their censoring, either at study completion or prematurely as drop-out.
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Overall Group
Number analyzed (Participants) | 1395
Cases per 100 person-years
  All subjects | 3.63 [3.12 to 4.20]
  Non-case: number analyzed (Participants) | 1269
  Non-case | 3.13 [2.64 to 3.69]
  WHO RSV LRTI: number analyzed (Participants) | 126
  WHO RSV LRTI | 9.44 [6.65 to 13.01]

ADVERSE EVENTS:
Time Frame: No adverse events were collected during this prospective epidemiological study.
Description: No adverse events were collected during this prospective epidemiological study; blood sampling was the only invasive procedure done to assess the disease burden of RSV associated, suspected LRTIs and incidence of wheeze and asthma.
Arm/Group | Overall Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT01995175/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT01995175/SAP_001.pdf